CLINICAL TRIAL: NCT06811311
Title: Neurophysiological and Psychological Effects of Ericksonian Hypnotherapy on Generalized Anxiety Disorder: An EEG-Based Clinical Study
Brief Title: EEG Study on Neurophysiological and Psychological Effects of Ericksonian Hypnotherapy in Generalized Anxiety Disorder
Acronym: EEG-HypnoGAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Collaborators: Istanbul Nisantasi University (Other); Beykoz University (Other)
Responsible Party: Principal Investigator, Selami Varol Ülker, Dr, Uskudar University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uskudar University EEG
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Generalized Anxiety Disorder (GAD); Anxiety Disorders; Psychophysiological Disorders; Stress-Related Disorders
Keywords: Ericksonian Hypnotherapy; Hypnosis and Anxiety; EEG Neurophysiology; Anxiety Treatment; Cognitive-Emotional Regulation
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders; Psychophysiologic Disorders

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled clinical trial with two parallel groups: one receiving Ericksonian hypnotherapy and the other serving as a no-treatment control group. The study examines changes in neurophysiological (EEG) and psychological (anxiety severity, emotion regulation, quality of life) parameters before and after treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ericksonian Hypnotherapy Group (Experimental): Participants in this group will receive 12 individual Ericksonian hypnotherapy sessions, each lasting 90 minutes, over a 12-week period. The hypnotherapy will be delivered by trained clinicians and will incorporate permissive language, metaphorical storytelling, and indirect suggestions tailored to address cognitive and emotional patterns associated with Generalized Anxiety Disorder.
  Interventions: Behavioral: Ericksonian Hypnotherapy
- Control Group (No Intervention): Participants in this group will receive no psychological intervention during the study period. They will continue their usual daily routines without structured psychotherapy, hypnosis, or additional psychological treatment. They will complete baseline and post-study assessments without receiving active treatment.

INTERVENTIONS:
Behavioral: Ericksonian Hypnotherapy — Ericksonian hypnotherapy is a therapeutic approach that utilizes indirect suggestion, storytelling, and metaphorical language to induce a trance state and facilitate psychological change. This intervention aims to reduce anxiety symptoms, improve emotional regulation, and alter neurophysiological responses as measured by EEG. Participants will undergo 12 individual sessions, each lasting 90 minutes, over a period of 12 weeks.
  Arms: Ericksonian Hypnotherapy Group

SUMMARY:
This study examines the neurophysiological and psychological effects of Ericksonian hypnotherapy in individuals diagnosed with Generalized Anxiety Disorder (GAD). Using electroencephalography (EEG), the study aims to assess changes in brain activity and anxiety symptoms before and after treatment.

A total of 60 participants will be recruited from both governmental and private psychiatric clinics in Istanbul. Participants will be randomly assigned to either the intervention group (receiving 12 Ericksonian hypnotherapy sessions over 12 weeks) or the control group (receiving no intervention).

The primary outcome measures include changes in EEG patterns, specifically alpha, theta, and frontal asymmetry indices, and changes in anxiety severity, measured by the Beck Anxiety Inventory (BAI), Generalized Anxiety Disorder-7 (GAD-7), and State-Trait Anxiety Inventory (STAI). Secondary measures include emotional regulation (DERS) and quality of life (WHOQOL-BREF).

This study aims to provide scientific evidence on the effectiveness of Ericksonian hypnotherapy as a complementary treatment for GAD and its impact on brain function and emotional well-being.

DETAILED DESCRIPTION:
This study investigates the neurophysiological and psychological effects of Ericksonian hypnotherapy in individuals diagnosed with Generalized Anxiety Disorder (GAD) using electroencephalography (EEG). The research aims to determine whether Ericksonian hypnotherapy produces measurable changes in brain activity and anxiety symptoms.

A total of 60 participants (30 per group) will be recruited from both governmental and private psychiatric clinics in Istanbul. Participants will be diagnosed with GAD based on DSM-5 criteria and will undergo structured psychiatric evaluation before inclusion.

Study Design Intervention Group (n = 30): Participants will receive 12 individual Ericksonian hypnotherapy sessions, each lasting 90 minutes, delivered over 12 weeks. The hypnotherapy protocol will include permissive language, metaphorical storytelling, and indirect suggestions tailored to anxiety-related cognitive and emotional patterns.

Control Group (n = 30): Participants will receive no psychological intervention during the study period.

Both groups will undergo baseline and post-intervention EEG measurements and complete psychological assessments.

Primary Outcome Measures:

EEG Changes: Resting-state and task-based EEG recordings will be analyzed for alpha, theta power, frontal asymmetry indices, and event-related potentials (ERPs: P300, N200) to assess neurophysiological effects of hypnotherapy.

Anxiety Severity: Beck Anxiety Inventory (BAI), Generalized Anxiety Disorder-7 (GAD-7), and State-Trait Anxiety Inventory (STAI) will be used to measure anxiety symptom changes.

Secondary Outcome Measures:

Emotional Regulation: Measured using the Difficulties in Emotion Regulation Scale (DERS).

Quality of Life: Evaluated with the World Health Organization Quality of Life Scale (WHOQOL-BREF).

Timeline:

Recruitment Period: February 1, 2025 - March 15, 2025 Baseline Assessments: March 2025 Intervention Period: April 1, 2025 - June 2025 Post-Intervention Assessments: July 2025 This study aims to provide scientific evidence on the efficacy of Ericksonian hypnotherapy as a complementary treatment for Generalized Anxiety Disorder by evaluating both neurophysiological and psychological changes. Findings may contribute to the development of alternative therapeutic approaches for anxiety disorders.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Generalized Anxiety Disorder (GAD) based on DSM-5 criteria
* Aged 18-65 years
* Capable of providing written informed consent
* Fluent in Turkish (for hypnosis and assessments)
* Not currently receiving psychotherapy or pharmacological treatment for anxiety

Exclusion Criteria:

* Presence of comorbid psychiatric disorders (e.g., schizophrenia, bipolar disorder, major depression requiring immediate intervention)
* History of neurological conditions (e.g., epilepsy, traumatic brain injury, stroke)
* Current use of medications affecting EEG activity (e.g., benzodiazepines, SSRIs, antipsychotics)
* Previous experience with hypnotherapy (to avoid expectancy bias)
* Substance abuse or dependence within the last six months
* Pregnancy or breastfeeding
* Severe medical conditions that may interfere with participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
EEG Changes in Brain Activity | Baseline (Pre-intervention) and Post-intervention (12 weeks)
  Measure: Changes in alpha, theta power, and frontal asymmetry indices before and after intervention Description: EEG will be used to assess changes in resting-state brain activity and event-related potentials (ERPs: P300, N200), evaluating neurophysiological effects of Ericksonian hypnotherapy.
Beck Anxiety Inventory (BAI) | Baseline and Post-intervention (12 weeks)
  Change in BAI scores (0-63, higher scores indicate more severe anxiety).

SECONDARY OUTCOMES:
Generalized Anxiety Severity (Generalized Anxiety Disorder-7, GAD-7) | Baseline and Post-intervention (12 weeks)
  Change in GAD-7 scores (0-21, higher scores indicate more severe anxiety)
State and Trait Anxiety Levels (State-Trait Anxiety Inventory, STAI) | Baseline and Post-intervention (12 weeks)
  Change in STAI scores (20-80, higher scores indicate greater anxiety).
Difficulties in Emotion Regulation Scale, (DERS) | Baseline and Post-intervention (12 weeks)
  Change in DERS scores (36-180, higher scores indicate greater emotion regulation difficulties).
World Health Organization Quality of Life Scale, (WHOQOL-BREF) | Baseline and Post-intervention (12 weeks)
  Change in WHOQOL-BREF scores (0-100, higher scores indicate better quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Selami Varol Ülker, Phd, Principal Investigator — Üsküdar University; Metin Çınaroğlu, Phd, Principal Investigator — Istanbul Nisantasi University
Locations (1):
- Üsküdar University, Neuro-Psychology Lab, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified EEG data and psychological assessment scores will be shared with qualified researchers upon reasonable request. Data will be made available after study completion and publication of results, following approval by the ethics committee. Data access will be granted through a secure repository or institutional agreement.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: After the results will be published in a peer review SSCI indexed journal
Access Criteria: Access to de-identified EEG and psychological assessment data will be granted to qualified researchers affiliated with recognized academic institutions or research organizations. Researchers must submit a formal data request, including a research proposal, to the study's principal investigator. Approved requests will receive access via a secure repository or institutional agreement, subject to ethical and data protection compliance.